CLINICAL TRIAL: NCT03639818
Title: COGSTIM 2 Study: Management by Individual Cognitive Remediation of Cognitive Disorders of HIV Infected Patients Controlled by Antiretroviral Treatment
Brief Title: Management by Individual Cognitive Remediation of Cognitive Disorders of HIV Infected Patients
Acronym: COGSTIM2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-15
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): HIV patients
  Interventions: Other: individual sessions of cognitive remediation

INTERVENTIONS:
Other: individual sessions of cognitive remediation — The cognitive remediation will be led by a psychologist specialized in neuropsychology, trained and experienced in this method. Cognitive remediation will be performed at a rate of 1 to 2 sessions per week for the duration of the study. This treatment will be carried out individually for half in face-to-face session in the clinical immuno-hematology department, face-to-face with the neuropsychologist, half at home with computer-based home exercises using PRESCO software ® from HAPPYNEURON®

SUMMARY:
Despite sustained inhibition of viral replication in plasma undergoing treatment, nearly 30% of HIV-infected patients have HIV-related cognitive impairment. To date, no therapeutic strategy has demonstrated clinical efficacy. The initial hypothesis is to use the non-medical techniques of cognitive remediation commonly practiced in the treatment of Alzheimer's disease to allow improvement or even regression of cognitive disorders in HIV-infected people (PHAs) who are virologically tested on antiretroviral combination therapy (ART). Some recent pilot studies using individual computer-based cognitive remediation strategies show improved test performance. However, none have studied the impact of this strategy on PPHIV with cognitive impairment.

A single-center pilot study evaluating the efficacy of an individual cognitive remediation program for 6 months on the improvement of cognitive impairment in patients with stable plasma HIV viral load that is undetectable under stable antiretroviral combination (cART) cognitive disorders related to HIV infection.

The primary objective is to demonstrate improvement through a 6-month individual cognitive remediation program on cognitive impairment (1 standard deviation variations on 2 M6 neuropsychological tests) in controlled HIV-positive individuals under cART with cognitive disorders related to HIV.

Methodology: Monocentric, prospective, pilot study of 40 patients performed in an open period of 25 months. The inclusion period is 13 months and the participation duration per patient is 12 months. After an inclusion visit, patients start 15 days of individual cognitive remediation sessions. The cognitive remediation will be led by a psychologist specialized in neuropsychology, trained and experienced in this method. Cognitive remediation will be performed at a rate of 1 to 2 sessions per week. Each patient will be assessed initially (M0) at 6 months (M6) and 12 months (M12: 6 months after stopping cognitive remediation) with a battery of standardized neuropsychological (NP) tests performed by a neuropsychologist.

Primary endpoint: Improved cognitive impairment after 6 months of cognitive remediation, with each patient being their own control, defined by improvement on at least 2 tests of 1 standard deviation minimum.

DETAILED DESCRIPTION:
Background: Despite sustained inhibition of viral replication in plasma undergoing treatment, nearly 30% of HIV-infected patients have HIV-related cognitive impairment. To date, no therapeutic strategy has demonstrated clinical efficacy. The initial hypothesis is to use the non-medical techniques of cognitive remediation commonly practiced in the treatment of Alzheimer's disease or traumatic brain injury to allow improvement or even regression of cognitive disorders in HIV-infected people (PHAs) who are virologically tested on antiretroviral combination therapy (ART). If this hypothesis is validated, this study will develop additional care structures and / or skills for the management of these cognitive disorders. Some recent pilot studies using individual computer-based cognitive remediation strategies show improved test performance. However, none have studied the impact of this strategy on PPHIV with cognitive impairment.

Study description: A single-center pilot study evaluating the efficacy of an individual cognitive remediation program for 6 months on the improvement of cognitive impairment in patients with stable plasma HIV viral load that is undetectable under stable antiretroviral combination (cART). cognitive disorders related to HIV infection. Cognitive remediation will be based on individual face-to-face cognitive remediation sessions with a neuropsychologist and on patients with severe psychiatric conditions or treatments that may interfere with neuropsychological (NP) testing. this search.

Main Objective: The primary objective is to demonstrate improvement through a 6-month individual cognitive remediation program on cognitive impairment (1 standard deviation variations on 2 M6 neuropsychological tests) in controlled HIV-positive individuals under cART with cognitive disorders related to HIV.

Secondary objectives:

1. Analyze the evolution of cognitive disorders 6 months after stopping cognitive remediation,
2. To analyze the evolution of the cognitive disorders in the cases of a duration of the remediation inferior to 6 months and superior to 2 months
3. Determine the most sensitive psychometric tests among those screened for asymptomatic and minor cognitive impairment in the HIV patient
4. Evaluate the impact of these therapeutic treatments on the quality of life, social autonomy and self-esteem
5. Characterize cognitive impairment in HIV patients according to Frascatti criteria, Glissen criteria and norms routinely used in neuropsychology routinely for each test
6. Describe the risk factors and co-morbidities associated with cognitive impairment

Methodology: Monocentric, prospective, pilot study of 40 patients performed in an open period of 25 months. The inclusion period is 13 months and the participation duration per patient is 12 months. After an inclusion visit (inclusion and non-inclusion criteria checks, data collection, clinical examination, psychometric test battery, Beck's scale and STAI-Y for evaluation of anode-depressive symptoms), patients start 15 days of individual cognitive remediation sessions. The cognitive remediation will be led by a psychologist specialized in neuropsychology, trained and experienced in this method. Cognitive remediation will be performed at a rate of 1 to 2 sessions per week for the duration of the study. This treatment will be carried out individually for half in face-to-face session in the clinical immuno-hematology department, face-to-face with the neuropsychologist, half at home with computer-based home exercises using PRESCO software ® from HAPPYNEURON®. Each patient will be assessed initially (M0) at 6 months (M6) and 12 months (M12: 6 months after stopping cognitive remediation) with a battery of standardized neuropsychological (NP) tests performed by a neuropsychologist.

Primary endpoint: Improved cognitive impairment after 6 months of cognitive remediation, with each patient being their own control, defined by improvement on at least 2 tests of 1 standard deviation minimum.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive patient1
* With a plasma viral load below the detection threshold for 6 months minimum, with the exception of blips defined by the presence of a detectable viral load <1000 copies / ml undetectable controlled on another successive collection.
* Triple antiretroviral tritherapy stable for 6 months
* Presenting a cognitive disorder proven by an alteration of at least 2 of the cognitive fields evaluated by psychometric tests for 6 months minimum
* 18 years <age <65 years
* Absence of marked depression defined by Beck score <16 (Appendix 13)
* Affiliated to the social security system,

  -) Having signed the consent form.
* Having made a balance of cognitive disorders eliminating any other cause of cognitive disorders including at least a cerebral MRI or brain CT () injected)
* Familiar with the use of computer tools (Having computer equipment with an internet connection or accepting to come on site to use the software of cognitive remediation exercises)

Exclusion Criteria:

* Patient with a psychiatric pathology diagnosed and followed for more than 6 months that could interfere with the psychometric evaluation, with the exception of depression with Beck score> 16 on the inclusion report
* Patient with a poor understanding of French,
* Active addiction
* Alcohol dependence
* Patient under guardianship,
* Patient with HIV-related dementia
* Child B or C liver cirrhosis (Appendix 17)
* Severe renal insufficiency (Cockcroft clearance of creatinine <30 ml / min)
* Any severe clinical event in the opinion of the investigator that could interfere with the strategy under study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
number of cognitive disorders | 6 months
  Improvement of cognitive disorders after 6 months of cognitive remediation, each patient being his own control, defined by the improvement on at least 2 tests of 1 minimum standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, MD, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France